CLINICAL TRIAL: NCT06635655
Title: Evaluation of Medical Benefit of a New Prosthetic Leg Designed to Decrease Mental Workload in People With Lower Limb Amputation
Brief Title: Assessment of the Prosthetic System Impact on Mental Workload in Above-knee Lower Limb Amputees.
Acronym: INCREMENT
Status: Recruiting | Type: Observational
Sponsor: Proteor Group (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00581-44
Record Dates: First submitted 2024-10-04; First posted 2024-10-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: microprocessor controlled; lower limb prosthesis; mental workload
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New generation of lower limb prosthesis provide improved functionalities. They are usually studied in the scope of biomechanics, sometimes PROMs like quality of life. Following users feedback, it is desirable to better understand why and how mental workload is impacted by new technologies or features. This clinical investigation will try to measure a difference between different prosthetic systems, in lab and in daily life.

DETAILED DESCRIPTION:
Multicentric, national, observational, prospective study, using AB type SCED.

ELIGIBILITY:
Inclusion Criteria:

* above-knee lower limb amputation
* using an above-knee prosthesis with prosthetic knee and foot
* eligible to use Synsys
* able to design therapeutic objectives for the GAS
* having a smartphone

Exclusion Criteria:

* protected person
* pregnant or breast-feeding lady
* knee-to-ground height lower than 43cm
* weighting more than 125kg
* using their prosthesis for less than 2 weeks
* not covered by health insurance
* aged less than 18 or more than 84 years old
* bilateral amputee or hip disarticulated

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population usually living or receiving care around investigation centers
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale (GAS) | From enrollment to the end of treatment at 8 weeks
  Scale from -3 to +2. The higher the better.
  -3 being a deterioration, -2 being the baseline, 0 the objective, +2 the maximum

SECONDARY OUTCOMES:
L-test and Dual-task L-test | Initial visit, at 4 weeks, and at 8 weeks
  To assess locomotor capacity in divided attention on a short period
Two-minute walk test (2MWT) and 2MWT in divided attention | Initial visit, at 4 weeks, and at 8 weeks
  to assess locomoto capacity and mental worload during a 2-minute exercise
Activity Balance Confidence Scale (ABC-scale) | at 4 weeks, and at 8 weeks
  Patient reported balance confidence Scale from 0% (minimum) to 100% (maximum), the higher the better.
Prosthesis Evaluation Questionnaire (PEQ-A) | at 4 weeks, and at 8 weeks
  Patient reported satisfaction Visual Analog Scale from 0% (minimum) to 100% (maximum) The higher the better
Stumbles and falls | at 4 weeks, and at 8 weeks
  Self-reported number The lower the better

CONTACTS AND LOCATIONS:
Overall Officials: Laurine Calistri, MS, Study Director — Proteor Group; Isabelle Loiret, DR, Principal Investigator — UGECM Nord-Est, IRR, Centre Louis Pierquin
Locations (1):
- Multiple sites, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: Undecided